CLINICAL TRIAL: NCT01254552
Title: Assessment With Cardiac Computed Tomography Angiography (CCTA) and Magnetic Resonance Imaging (MRI) in Asymptomatic Patients With Type 2 Diabetes for Detection of Unrecognized Myocardial Scar in Subclinical Coronary Atherosclerosis
Brief Title: Assessment With CCTA and MRI in Asymptomatic Patients With Type 2 Diabetes for Detection of Unrecognized Myocardial Scar in Subclinical Coronary Atherosclerosis
Acronym: ACCREDIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISO-44-011
Record Dates: First submitted 2010-10-13; First posted 2010-12-06 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus; Coronary Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — iobitridol; gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dotarem and Xenetix 350 (Experimental)
  Interventions: Drug: iobitridol; Drug: gadoterate meglumine

INTERVENTIONS:
Drug: iobitridol — Xenetix 350 was administered at a dose up to 180 ml, according to the patient's body weight measured on the day of administration.
  Other Names: Xenetix
Drug: gadoterate meglumine — Dotarem was administered at a dose of 0.1 mmol/kg body weight (0.2 ml/kg body weight)
  Other Names: gadoteric acid; Dotarem

SUMMARY:
The study aimed to prospectively investigate the prevalence of myocardial scar on Dotarem-enhanced Cardiovascular Magnetic Resonance Imaging (MRI) in asymptomatic patients with type-2 Diabetes Mellitus and to assess its correlation with subclinical coronary artery disease on Cardiac Computed Tomography Angiography (CCTA).

DETAILED DESCRIPTION:
Patients underwent a cardiac MRI examination with Dotarem within 60 days after screening visit. The myocardial CCTA examination with Xenetix 350 was performed within 1 to 30 days (but no sooner than 24 hours) after the MRI examination.

ELIGIBILITY:
Inclusion Criteria:

* Patient with onset of type 2 diabetes occurred at age 30 years or older
* Patient between the ages of 50 and 75 years at enrolment time
* Patient with at least two identified cardiac risk factors who will undergo a CMR and a CCTA examinations to evaluate his/her coronary and cardiac status

Exclusion Criteria:

* Patient with angina pectoris or chest discomfort
* Patient with stress test or invasive coronary angiography within the prior 3 years
* Patient with history of myocardial infarction, overt non compensated heart failure, or coronary revascularization
* Patient with hemodynamic instability.
* Patient with a contraindication or intolerance to Beta-Blocker administration

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Dotarem and Xenetix 350: All patients were planned to undergo a MRI examination with Dotarem and a myocardial CCTA examination with Xenetix 350 to evaluate his/her coronary and cardiac status.
Period: Screening Visit
Arm/Group | Dotarem and Xenetix 350
Started | 351
Completed | 348
Not Completed | 3
Period: Delayed-enhanced MRI With Dotarem
Arm/Group | Dotarem and Xenetix 350
Started | 348
Completed | 328
Not Completed | 20
Period: CCTA With Xenetix 350
Arm/Group | Dotarem and Xenetix 350
Started | 328
Completed | 322
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- All Included Patients: All patients included in the study.
Arm/Group | All Included Patients
Number analyzed (Participants) | 348
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.18 (6.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212
  Male | 136

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Occult Myocardial Scar on Delayed-enhanced MRI in Asymptomatic Patients With Type 2 Diabetes Mellitus
Time Frame: From 1 week to 2 months (after the collection of data corresponding to cardiac MRI and CCTA examinations)
Measure: Count of Participants; unit: Participants
Groups:
- Intention To Treat Population: All patients with a valid MRI and CCTA examinations.
Arm/Group | Intention To Treat Population
Number analyzed (Participants) | 322
Participants | 23
Statistical Analysis 1: Comparison: Intention To Treat Population; Test type: Other; rate = 0.071, 95% CI 2-sided [0.043 to 0.100]

2. Secondary Outcome: Number of Patients With and Without Occult Myocardial Scar on Cardiac MRI According to the Degree of Stenosis
Description: The degree of coronary artery stenosis on CCTA was assessed according to the following scale:
  * No stenosis: 0%
  * Non significant stenosis: 1-50%
  * Significant stenosis >50% and ≤99%
  * Occlusion: 100%
Time Frame: From 1 week to 2 months (after the collection of data corresponding to cardiac MRI and CCTA examinations)
Measure: Count of Participants; unit: Participants
Groups:
- Patients Without Occult Myocardial Scar: Patients without Occult Myocardial Scar on cardiac MRI
- Patients With at Least One Occult Myocardial Scar: Patients with at least one Occult Myocardial Scar on cardiac MRI
Arm/Group | Patients Without Occult Myocardial Scar | Patients With at Least One Occult Myocardial Scar
Number analyzed (Participants) | 299 | 23
Participants
  No stenosis: 0% | 80 | 2
  Non-significant stenosis: 1-50% | 152 | 8
  Significant stenosis: >50% and ≤99% | 61 | 12
  Occlusion: 100% | 6 | 1

ADVERSE EVENTS:
Time Frame: From the signature of the informed consent form until 30 minutes after the end of CCTA examination i.e. from 2 days to 3 months
Description: The analysis of adverse events was performed on the safety population that includes all patients receiving at least one injection of contrast agent regardless of the quantity. Post-injection AEs collected between Dotarem and Xenetix 350 injection, during Xenetix 350 injection and after Xenetix 350 injection are presented.
Groups:
- Between Dotarem and Xenetix 350 Injection: Adverse events that occurred after Dotarem injection (MRI examination) and before Xenetix 350 injection (CCTA examination)
- During Xenetix 350 Injection: Adverse events that occurred during injection of Xenetix 350 (CCTA examination)
- After Xenetix 350 Injection: Adverse events that occurred after the injection of Xenetix 350 (CCTA examination)
Arm/Group | Between Dotarem and Xenetix 350 Injection | During Xenetix 350 Injection | After Xenetix 350 Injection
All-Cause Mortality (participants affected / at risk) | 0/328 | 0/328 | 0/328
Serious Adverse Events (participants affected / at risk) | 0/328 | 0/328 | 0/328
Other Adverse Events (participants affected / at risk) | 8/328 | 12/328 | 7/328
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Between Dotarem and Xenetix 350 Injection (N=328) | During Xenetix 350 Injection (N=328) | After Xenetix 350 Injection (N=328)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other